CLINICAL TRIAL: NCT04445337
Title: Stellate Ganglion Blockade in COVID-19 Positive Patients
Brief Title: Stellate Ganglion Blockade in Corona Virus 2019 (COVID-19) Positive Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to recruit sufficient number of subjects.
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0523-20-FB
Record Dates: First submitted 2020-06-09; First posted 2020-06-24 (Actual); Results first posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-12

CONDITIONS: COVID 19; ARDS
Keywords: stellate ganglion; perineural block
MeSH Terms: conditions — COVID-19 | interventions — Clonidine; Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: Open-label use of stellate ganglion block.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Open Label SGB (Experimental): Initial perineural bolus injection - clonidine 100 mcg, Decadron PF 5mg, and 0.25% bupivacaine 5 ml will be used for SGB block.
  Interventions: Drug: Stellate Ganglion Block
- Control Arm (No Intervention): There will be no sham procedure for the control group. The control group will have nitric oxide levels performed once a day by a member of the research team. Lab draws will be drawn at the same frequency as the treatment group.

INTERVENTIONS:
Drug: Stellate Ganglion Block — An injection of local anesthetic into the front of the neck. SGB involves placing a small tube into the front of your neck, toward nerves at the back of your neck. This is done with the help of an x-ray machine or ultrasound device. The tube is left in place so you can get medication thru it for five days. Then the tube is taken out.
  The medication used for the block are clonidine 100 mcg, Decadron PF 5mg and 0.25% bupivacaine 5 mL. This medication will be administered once during the block. These medications are approved by the Food and Drug Administration (FDA).
  Other Names: Catapres, Decadron & Marcaine administration
  Arms: Open Label SGB

SUMMARY:
This study will establish the safety and efficacy of using stellate ganglion blocks in patients with acute respiratory distress syndrome (ARDS) due to COVID-19 disease.

DETAILED DESCRIPTION:
The stellate ganglion block (SGB) will be performed in the ICU. Nurse will provide patient monitoring and assistance during the procedure. Standard monitors and advanced cardiovascular life support (ACLS) resuscitative equipment will be immediately available. A norepinephrine solution will be at bedside to treat potential hypotension associated with SGB. The SGB perineural catheter will be placed using standard sterile technique. Initial perineural bolus injection - clonidine 100 mcg, Decadron sodium phosphate (PF) 5mg, and 0.25% bupivacaine 5 ml is delivered. An ONQ brand perineural infusion 0.2% bupivacaine will be initiated at 2ml/hr for 5 days. Acute pain service will discontinue infusion and remove the catheter after 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Any patient between the ages of 19-85 with laboratory established COVID-19 infection via Real-Time Reverse Transcription-Polymerase Chain Reaction (rRT-PCR) requiring critical care in an intensive care unit.
* Signs or symptoms consistent with ARDS must be present.
* The syndrome must present acutely, ratio of arterial oxygen partial pressure to fractional inspired oxygen (PaO2/FIO2) ≤ 200 mm Hg, bilateral infiltrates on chest radiograph or CT not due to cardiac failure, need for non-invasive or invasive mechanical ventilation, and any cardiac dysrhythmia (excluding sinus tachycardia).

Exclusion Criteria:

* Hemodynamic instability (>2 vasopressors)
* pre-hospital diagnosis of heart failure or fluid overload
* anatomical inability to perform block
* prior sympathectomy
* patient currently enrolled in another clinical trial for COVID-19 or respiratory distress/acute respiratory distress syndrome (ARDS)
* uncorrectable coagulopathy, already on Extracorporeal membrane oxygenation (ECMO), already on Nitric Oxide, pre-existing multi-organ failure (>2 organ systems).

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lankhorst, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label SGB: Initial perineural bolus injection - clonidine 100 mcg, Decadron sodium phosphate (PF) 5mg, and 0.25% bupivacaine 5 ml will be used for SGB block.
  Stellate Ganglion Block: An injection of local anesthetic into the front of the neck. Medication used for the block include- clonidine 100 mcg, Decadron PF 5mg, and 0.25% bupivacaine 5 ml is delivered.
- Control Arm: There will be no sham procedure for the control group. The control group will have nitric oxide levels performed once a day by a member of the research team. Lab draws will be drawn at the same frequency as the treatment group.
  Control: Standard of care. Observation.
Period: Overall Study
Arm/Group | Open Label SGB | Control Arm
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The enrollment was difficult and the data is insignificant and will not be useful to perform an analysis.
Groups:
- Stellate Ganglion Block: Initial perineural bolus injection - clonidine 100 mcg, Decadron PF 5mg, and 0.25% bupivacaine 5 ml will be used for SGB block.
  Stellate Ganglion Block: An injection of local anesthetic into the front of the neck. Medication used for the block include- clonidine 100 mcg, Decadron PF 5mg, and 0.25% bupivacaine 5 ml is delivered.
- Standard of Care: There will be no sham procedure for the control group. The control group will have nitric oxide levels performed once a day by a member of the research team. Lab draws will be drawn at the same frequency as the treatment group.
  Control: Standard of care. Observation.
- Total: Total of all reporting groups
Arm/Group | Stellate Ganglion Block | Standard of Care | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] |  | 50 [50 to 50] | 50 [50 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Safety of a New Modified Stellate Ganglia Block (SGB) in Acute Respiratory Distress Syndrome (ARDS)
Description: a) differences in mean/median values for SGB vs standard of care (SOC) will be assessed at each of the study designated time points for all the continuous biomarker measures - by assessing magnitude of difference and its 95% confidence level and testing differences for statistical significance at each of the time points;
Time Frame: 3 month
Population: Differences in mean/median values for SGB vs standard of care (SOC) will be assessed at each of the study designated time points for all the continuous biomarker measures - by assessing the magnitude of difference and its 95% confidence level and testing differences for statistical significance at each of the time points; Unable to recruit sufficient subjects. Only one subject was randomized to the control group and did not receive the intervention.
Groups:
- Open Label SGB: Initial perineural bolus injection - clonidine 100 mcg, Decadron PF 5mg, and 0.25% bupivacaine 5 ml will be used for SGB block.
  Stellate Ganglion Block: An injection of local anesthetic into the front of the neck. Medication used for the block include- clonidine 100 mcg, Decadron PF 5mg, and 0.25% bupivacaine 5 ml is delivered.
Arm/Group | Open Label SGB | Control Arm
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Evaluating Stellate Ganglion Block Adverse Events.
Description: e) Differences between SGB vs SOC in frequency and time to occurrence of cardiac arrhythmias;
Time Frame: 3 month
Population: Secondary outcome e) Differences between SGB vs SOC in frequency and time to occurrence of cardiac arrhythmias. Unable to recruit sufficient subjects. Only one subject was randomized to the control group and did not receive the intervention.
Arm/Group | Open Label SGB | Control Arm
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: There were no subjects in the intervention arm. Therefore the number of participants at risk was zero.
Arm/Group | Open Label SGB | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

LIMITATIONS AND CAVEATS:
Unable to recruit sufficient subjects. Only one subject was randomized to the control group and did not receive the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/37/NCT04445337/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT04445337/ICF_001.pdf